CLINICAL TRIAL: NCT00585065
Title: Cardiac Resynchronization Therapy for Children and Adolescents With Advanced Hearth Failure: A Pilot Study
Brief Title: CRT Pilot Study for Children With Heart Failure
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: 00015291
Record Dates: First submitted 2007-12-21; First posted 2008-01-03 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2021-04

CONDITIONS: Chronic Pediatric Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Pediatric and adolescent patients receiving CRT with BVP for treating chronic heart failure: Pediatric and adolescent patients who are receiving cardiac resynchronization therapy with biventricular pacing as a method of treating chronic heart failure. Children of both genders, who are followed in the Division of Pediatric Cardiology at Primary Children's Medical Center, who meet all inclusion and no exclusion criteria are eligible for participation in this clinical study.
  No intervention is administered as part of this study. Prospective longitudinal case series study to describe and evaluate clinical and hemodynamic effects of CRT and to identify echocardiographic predictors of positive response to CRT in Group described.
  Interventions: Device: CRT device implant

INTERVENTIONS:
Device: CRT device implant — The purpose of this study is to collect information on patients with chronic heart failure who have already been identified by their physician as candidates for CRT. All tests, including device implantation are standard of care for patients undergoing CRT. The only test involved in this study that is not standard of care is the quality of life questionnaire. Patients who undergo CRT system implant will be followed post-implant (up to 1 week), and at one month, three months, six months and twelve months. The only test involved in this study that is not standard of care is the quality of life questionnaire.

SUMMARY:
To collect information on pediatric patients receiving Cardiac Resynchronization Therapy (CRT) with permanent biventricular pacing (BVP) as a method of treating chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic and severe heart failure, NYHA class III or IV
2. Patients optimized and stable on diuretics and afterload reducing agents (with or without inotropes) for at least 1 week prior to enrollment
3. Chronic systemic ventricular dysfunction as defined in the protocol.
4. Intra ventricular conduction delay defined by spontaneous QRS duration > ULN for age.
5. All children from 1 to 18 years of age, both male and female, and all ethnic backgrounds.
6. Signed and dated informed consent.
7. Able to receive pectoral or abdominal implant.

Exclusion criteria:

1. Suspected acute myocarditis.
2. Significant ventricular dysfunction, secondary to acquired or congenital heart defects amenable to surgical correction.
3. Acute coronary syndrome.
4. Adolescents who are pregnant.
5. Patient with BVP device implanted previously.
6. Patient has had prior/past heart transplantation.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2006-01; Primary Completion 2008-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Collection of quality of life information using the Pediatric Quality of Life Inventory 4.0 (PedsQl v4.0) in children and adolescents with chronic, advanced heart failure (defined by NYHA Functional Classification). | Within 30 days of CRT implant to 12 months post implant
  Composed of 23 items comprising 4 dimensions. 5-point Likert scale from: 0 (Never) to 4 (Almost always).
  Higher scores = Better health related quality of life (HRQOL)
Collection of survival information using the Pediatric Quality of Life Inventory 4.0 (PedsQl v4.0) in children and adolescents with chronic, advanced heart failure (defined by NYHA Functional Classification). | Within 30 days of CRT implant to 12 months post implant
  Composed of 23 items comprising 4 dimensions. 5-point Likert scale from: 0 (Never) to 4 (Almost always).
  Higher scores = Better health related quality of life (HRQOL)

SECONDARY OUTCOMES:
Echocardiographic measurement predictors of positive response to cardiac resynchronization therapy (CRT) in children and adolescent patients according to the American Society of Echocardiography guidelines | Within 30 days of CRT implant to 12 months post implant
  Describe the relationship between echocardiographic measures and subject response to CRT

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Saarel, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States